CLINICAL TRIAL: NCT00699907
Title: A Prospective, Phase IIA Study of the Effect of Flutamide (125 MG/DAY) Taken for 6 Weeks on Expression of Potential Biomarkers of Flutamide Action in the Ovaries of Women at Increased Risk for Ovarian Cancer
Brief Title: Effect of Flutamide on Biomarkers in Blood and Tissue Samples From Patients at High Risk of Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04-0707-04; P30CA023074 (NIH)
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2017-12

CONDITIONS: Ovarian Cancer
Keywords: Ovarian epithelial cancer; High risk; Biomarkers
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Flutamide; Salicylic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Arm (Active Comparator): Patients received oral flutamide (125 MG) once daily for 6 weeks in the absence of unacceptable toxicity. Patients then underwent risk-reducing salpingo-oophorectomy.
  Interventions: Drug: flutamide
- High Risk Arm (No Intervention): High risk patients underwent risk-reducing salpingo-oophorectomy.
- Low Risk Arm (No Intervention): Low risk patients underwent salpingo-oophorectomy for a medical indication.

INTERVENTIONS:
Drug: flutamide — Patients receive oral flutamide (125 MG/DAY) once daily for 6 weeks in the absence of unacceptable toxicity.
  Other Names: Eulexin; Cytomid; Cebatrol; Chimax; Drogenil; Flucinom; Flutamin; Fugerel; Niftolide; Sebatrol
  Arms: Treatment Arm

SUMMARY:
Studying samples of blood and tissue in the laboratory from patients with a high risk of developing ovarian cancer may help doctors identify and learn more about biomarkers related to cancer. We hypothesized that (i) preclinical biologic evidence exists for the role of androgens in ovarian cancer development and (ii) flutamide treatment of women at high risk for ovarian cancer may identify meaningful tissue biomarkers of androgen action and of ovarian cancer initiation. This phase II trial studied the effect of flutamide on biomarkers in blood and tissue samples from patients at high risk of ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVE: Compare the biomarkers of patients at high risk for ovarian cancer who are undergoing prophylactic oophorectomy and are interested in taking flutamide vs patients at high risk for ovarian cancer who are undergoing prophylactic oophorectomy and are not interested in taking flutamide (control) vs patients who are undergoing oophorectomy for a medical indication (control).

OUTLINE: Patients who elected not to receive flutamide received prophylactic oophorectomy or oophorectomy for a medical indication. Patients who elected to receive flutamide received 125mg once daily for 6 weeks in the absence of unacceptable toxicity. Patients then underwent prophylactic oophorectomy. All patients underwent blood and ovarian tissue sample collection at the time of surgery for biomarker laboratory studies. Proteomic, microarray, and polymorphism analysis were performed on the blood and tissue samples.

ELIGIBILITY:
Inclusion Criteria for all patients:

* ≥ 18 years of age
* Able to comply with study and follow-up requirements

Inclusion Criteria for high risk patients:

* elected to undergo prophylactic salpingo-oophorectomy
* fertile patients must use effective non-hormonal contraception
* agreed to use a nonhormonal means of contraception before surgery
* serum bilirubin ≤ 1.0 x Upper Limit Normal (ULN), alkaline phosphatase, Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT) ≤ 2.5 x ULN
* serum creatinine ≤ 1.5 x ULN
* granulocyte count ≥ 1500/μL
* platelet count ≥ 75,000/μL
* hemoglobin ≥ 9 g/dL
* adequate complete blood count
* At high risk for developing ovarian cancer, as defined by any of the following:
* Breast Cancer carried a BRCA1 or BRCA2 deleterious mutation, a Lynch syndrome mutation, and/or defined by a family history of: 1 first-degree relative with epithelial ovarian cancer, ≥1 first-degree female relative with breast cancer when ≤40 years old, ≥1 first-degree female relative with breast cancer when ≤50 years old, male relative with breast cancer, and/or family history of breast cancer or ovarian cancer.

Inclusion Criteria for low risk patients:

* planning to undergo oophorectomy for a medical indication
* did not fulfill criteria for high risk of developing ovarian cancer

Exclusion criteria:

* liver disease, current alcohol abuse, or cirrhosis
* pregnancy or lactation
* current use of hormone therapy
* active treatment for cancer
* recent, current, or planned participation in another experimental drug study
* breast cancer within the past 5 years
* significant traumatic injury within the past 6 months
* major surgery within the past 6 months
* any disease, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that contraindicates the continued use of an investigational drug or that may render the patient at high risk from treatment complication

Ages: 18 Years to 83 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2005-01; Primary Completion 2012-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Setsuko K. Chambers, MD, Principal Investigator — University of Arizona Arizona Cancer Center
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gruessner C, Gruessner A, Glaser K, AbuShahin N, Zhou Y, Laughren C, Wright H, Pinkerton S, Yi X, Stoffer J, Azodi M, Zheng W, Chambers SK. Flutamide and biomarkers in women at high risk for ovarian cancer: preclinical and clinical evidence. Cancer Prev Res (Phila). 2014 Sep;7(9):896-905. doi: 10.1158/1940-6207.CAPR-13-0408. Epub 2014 Jun 20. PMID 24950779
- See also: American Journal of Cancer Research, 2014. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3902233/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the medical clinic prior to oophorectomy. Participants were recruited from January 2007 until June 2011.
Pre-assignment Details: Participants were assigned to groups immediately after being enrolled.
Period: Overall Study
Arm/Group | Treatment Arm | High Risk Arm | Low Risk Arm
Started | 14 | 57 | 56
Completed | 12 | 47 | 48
Not Completed | 2 | 10 | 8
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — No usable sample | 0 | 9 | 8

BASELINE CHARACTERISTICS:
Population: The Overall Number of Participants Analyzed represents all participants with a modified Histo-score that could be evaluated
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | High Risk Arm | Low Risk Arm | Total
Number analyzed (Participants) | 12 | 47 | 48 | 107
Age, Continuous [Mean (Full Range); unit: years] | 45.2 [36 to 58] | 46.9 [27 to 66] | 51.7 [21 to 81] | 48.9 [21 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 47 | 48 | 107
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 47 | 48 | 107

OUTCOME MEASURES:

1. Primary Outcome: Colony Stimulating Factor (CSF-1) Expression in Ovarian Endosalpingiosis
Description: CSF-1 levels were measured by immunohistochemistry (IHC).
  The modified H-Score assess extent of nuclear immunoreactivity applicable to steroid receptors.
  The modified H-scores total range is 0-300. A lower modified H-score indicates weakly staining nuclei. A higher modified H-score indicated strongly staining nuclei.
  This applies to all measures.
Time Frame: Surgery
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Modified H-Score
Arm/Group | Treatment Arm | High Risk Arm | Low Risk Arm
Number analyzed (Participants) | 7 | 24 | 15
Modified H-Score | 5 [0 to 210] | 130 [0 to 300] | 50 [5 to 270]
Statistical Analysis 1: Comparison: Treatment Arm vs High Risk Arm; Test type: Superiority or Other; p = 0.012, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: High Risk Arm vs Low Risk Arm; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test

2. Primary Outcome: Colony Stimulating Factor (CSF-1) Expression in Ovarian Epithelium
Description: CSF-1 levels were measured by immunohistochemistry (IHC).
Time Frame: Surgery
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Histo-score (H-Score)
Arm/Group | Treatment Arm | High Risk Arm | Low Risk Arm
Number analyzed (Participants) | 8 | 42 | 39
Histo-score (H-Score) | 0 [0 to 30] | 50 [0 to 210] | 0 [0 to 120]
Statistical Analysis 1: Comparison: Treatment Arm vs High Risk Arm; Test type: Superiority or Other; p = 0.010, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: High Risk Arm vs Low Risk Arm; Test type: Superiority or Other; p = 0.005, Wilcoxon Rank Sum Test

3. Primary Outcome: Colony Stimulating Factor (CSF-1) Expression in Ovarian Stroma
Description: CSF-1 levels were measured by immunohistochemistry (IHC).
Time Frame: Surgery
Measure: Median (Full Range); unit: Histo-score (H-Score)
Arm/Group | Treatment Arm | High Risk Arm | Low Risk Arm
Number analyzed (Participants) | 11 | 45 | 43
Histo-score (H-Score) | 5 [0 to 80] | 40 [5 to 160] | 35 [5 to 180]
Statistical Analysis 1: Comparison: Treatment Arm vs High Risk Arm; Test type: Superiority or Other; p = 0.0006, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: High Risk Arm vs Low Risk Arm; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test

4. Primary Outcome: Colony Stimulating Factor-1 Receptor (CSF-1R) Expression in Ovarian Endosalpingiosis
Description: CSF-1R levels were measured by immunohistochemistry (IHC).
Time Frame: Surgery
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Histo-score (H-Score)
Arm/Group | Treatment Arm | High Risk Arm | Low Risk Arm
Number analyzed (Participants) | 6 | 21 | 16
Histo-score (H-Score) | 15 [0 to 60] | 160 [5 to 285] | 75 [5 to 195]
Statistical Analysis 1: Comparison: Treatment Arm vs High Risk Arm; Test type: Superiority or Other; p = 0.009, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: High Risk Arm vs Low Risk Arm; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test

5. Primary Outcome: Colony Stimulating Factor-1 Receptor (CSF-1R) Expression in Ovarian Epithelium
Description: CSF-1R levels were measured by immunohistochemistry (IHC).
Time Frame: Surgery
Measure: Median (Full Range); unit: Histo-score (H-Score)
Arm/Group | Treatment Arm | High Risk Arm | Low Risk Arm
Number analyzed (Participants) | 12 | 41 | 36
Histo-score (H-Score) | 0 [0 to 160] | 40 [0 to 270] | 20 [2 to 270]
Statistical Analysis 1: Comparison: Treatment Arm vs High Risk Arm; Test type: Superiority or Other; p = 0.037, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: High Risk Arm vs Low Risk Arm; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test

6. Primary Outcome: Colony Stimulating Factor-1 Receptor (CSF-1R) Expression in Ovarian Stroma
Description: CSF-1R levels were measured by immunohistochemistry (IHC).
Time Frame: Surgery
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Histo-score (H-Score)
Arm/Group | Treatment Arm | High Risk Arm | Low Risk Arm
Number analyzed (Participants) | 12 | 42 | 42
Histo-score (H-Score) | 20 [0 to 40] | 40 [0 to 210] | 53 [0 to 195]
Statistical Analysis 1: Comparison: Treatment Arm vs High Risk Arm; Test type: Superiority or Other; p = 0.010, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: High Risk Arm vs Low Risk Arm; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test

7. Primary Outcome: Tyrosine Kinase V-erb-b2 Erythroblastic Leukemia Viral Oncogene Homolog-4 (ErbB4) Expression in Ovarian Endosalpingiosis
Description: ErbB4 levels were measured by immunohistochemistry (IHC).
Time Frame: Surgery
Measure: Median (Full Range); unit: Histo-score (H-Score)
Arm/Group | Treatment Arm | High Risk Arm | Low Risk Arm
Number analyzed (Participants) | 7 | 19 | 9
Histo-score (H-Score) | 5 [0 to 30] | 60 [5 to 270] | 10 [5 to 270]
Statistical Analysis 1: Comparison: Treatment Arm vs High Risk Arm; Test type: Superiority or Other; p = 0.005, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: High Risk Arm vs Low Risk Arm; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test

8. Primary Outcome: Tyrosine Kinase V-erb-b2 Erythroblastic Leukemia Viral Oncogene Homolog-4 (ErbB4) Expression in Ovarian Epithelium
Description: ErbB4 levels were measured by immunohistochemistry (IHC).
Time Frame: Surgery
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Histo-score (H-Score)
Arm/Group | Treatment Arm | High Risk Arm | Low Risk Arm
Number analyzed (Participants) | 8 | 33 | 20
Histo-score (H-Score) | 0 [0 to 15] | 55 [0 to 270] | 0 [0 to 285]
Statistical Analysis 1: Comparison: Treatment Arm vs High Risk Arm; Test type: Superiority or Other; p = 0.006, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: High Risk Arm vs Low Risk Arm; Test type: Superiority or Other; p = 0.005, Wilcoxon Rank Sum Test

9. Primary Outcome: Tyrosine Kinase V-erb-b2 Erythroblastic Leukemia Viral Oncogene Homolog-4 (ErbB4) Expression in Ovarian Stroma
Description: ErbB4 levels were measured by immunohistochemistry (IHC).
Time Frame: Surgery
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Histo-score (H-Score)
Arm/Group | Treatment Arm | High Risk Arm | Low Risk Arm
Number analyzed (Participants) | 11 | 36 | 23
Histo-score (H-Score) | 10 [0 to 60] | 90 [10 to 285] | 30 [10 to 255]
Statistical Analysis 1: Comparison: Treatment Arm vs High Risk Arm; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: High Risk Arm vs Low Risk Arm; Test type: Superiority or Other; p = 0.005, Wilcoxon Rank Sum Test

ADVERSE EVENTS:
Arm/Group | Treatment Arm | High Risk Arm | Low Risk Arm
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 9/12 | 0/47 | 0/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=12) | High Risk Arm (N=47) | Low Risk Arm (N=48)
Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Endocrine (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Other (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urine color change (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal/Soft Tissue - other (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pain - Head/headache (General disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes